CLINICAL TRIAL: NCT04324346
Title: Evaluation of Central Venous Catheters Used for Chemotherapy in Women With Breast Cancer - An Interdisciplinary Randomized Controlled Study of Complications, Material Wear, Staff- and Patient Perspectives, and Health Economy.
Brief Title: Central Catheters Used for Chemotherapy in Women With Breast Cancer
Acronym: PICC&PAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish Red Cross University College (Other)
Collaborators: Karolinska Institutet (Other); KTH Royal Institute of Technology (Other); Karolinska University Hospital (Other); Stockholm South General Hospital (Other); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Gunilla Bjorling, Professor, Swedish Red Cross University College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: RKH2014.1
Record Dates: First submitted 2018-09-04; First posted 2020-03-27 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Catheter Related Complications
Keywords: picc-line; central venous access port; catheter related complications; Infections; thrombosis; Material degradation; Health economic costs; Bio-material; Health related quality of life
MeSH Terms: conditions — Infections; Thrombosis | interventions — Docetaxel; fluorescein isothiocyanate-keyhole limpet hemocyanin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PICC-Line (Experimental): Women allocated to PICC-line when receiving chemotherapy
  Interventions: Drug: FEC75 (or EC90) x 6; Drug: FEC100 + Taxotere (EC90 + Taxotere) 3+3; Drug: Paclitaxel
- Subcutaneous Venous Access Port (SVAP) (Experimental): Women allocated to SVAP when receiving chemotherapy
  Interventions: Drug: FEC75 (or EC90) x 6; Drug: FEC100 + Taxotere (EC90 + Taxotere) 3+3; Drug: Paclitaxel

INTERVENTIONS:
Drug: FEC75 (or EC90) x 6 — Type of Chemotherapy
Drug: FEC100 + Taxotere (EC90 + Taxotere) 3+3 — Type of Chemotherapy
Drug: Paclitaxel — Type of Chemotherapy

SUMMARY:
The overall aim of this study is to evaluate two different central venous lines, PICC-lines (PICC) and subcutaneous venous access ports (SVAP) used for chemotherapy in women with breast cancer. The study will compare complications, material wear of the catheters used, patients'- and health care professionals' experiences, and costs. The study will give knowledge about which central venous access that is the most advantageous regarding adjuvant chemotherapy for women with breast cancer in the aspects of safety, quality of care, and quality of life.

DETAILED DESCRIPTION:
N=250 women between 18 and 70 years of age with invasive breast cancer who are allocated to adjuvant or neo adjuvant chemotherapy during 18 weeks at the Department of Oncology at Karolinska University Hospital , Stockholm Sweden are eligible to participate in the present study. Exclusion criteria are cognitive dysfunction and/or inability to understand Swedish. Before participation an informed consent will be collected. The patients will be randomized to receive a PICC or a SVAP. Complications will be registered as well as the treatments.

Bacterial cultures will be taken at removal of PICC/SVAP. The used PICC/SVAP will be transported to the Royal Institute of Technology (KTH) and subjected to material analyses. Comparison with reference materials from the in-vitro study and with new reference catheters will be performed. Patient assessments with questionnaire concerning HRQL, illness perception, body imaging, life style and sleep disturbance will be collected at baseline and at the last chemotherapy session. Interviews with the patients about life situations will be conducted half through the chemotherapy treatment period.In- and out-patients costs, i.e. medication, materials, costs related to the care of the PICC/SVAP, costs for complications, additional costs for the patients regarding the treatment, etc., will be monitored and registered. In- and out-patient costs will also be monitored. Data from medical records concerning treatments for complications will also be taken into consideration.

ELIGIBILITY:
Inclusion Criteria:

* adjuvant or neo adjuvant chemotherapy,
* speak Swedish

Exclusion Criteria:

* cognitive dysfunction
* and/or inability to understand Swedish,
* recurrent breast cancer

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Complications | Through study completion up to 18 weeks
  all complications during the chemotherapy treatment period are registered

SECONDARY OUTCOMES:
Questionnaire EQ-5D | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  Health related quality of life is measured with scores and a scale using EQ-5D.
Questionnaire EORT-QLQ 30 | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  To measure Health related quality of life for patients with cancer the questionnaire EORT-QLQ 30 (Scores) is used.
Questionnaire EORT-QLQ BR32 | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  The Questionnaire EORT-QLQ BR32 (Scores) is used to measure Health related quality of life for patients with breast cancer
Questionnaire Insomnia Symptom Score | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  To measure Sleep disturbance the questionnaire Insomnia Symptom Score (Scores) is used.
Body Esteem Scale (BES) | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  The participants Body image is measured by Questionnaire: Body Esteem Scale (BES) (Scores)
Enriched Social Support Instrument (ESSI) | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  The participants social support is measured with the questionnaire: Enriched Social Support Instrument (ESSI) (Scores)
Brief-Illness Perception Questionnaire (B-IPQ) | At baseline, at 9 weeks and at end of treatment period 18 weeks (3 measurements)
  Illness Perception is measured with the questionnaire: Brief-Illness Perception Questionnaire (B-IPQ) (scores)

OTHER OUTCOMES:
Morphological material degradation | After study completion up to 18 weeks
  Morphological surface changes of PICC and SVAP after clinical use.
  End-ponits:
  • Material degradation of PICC/SVAP measured with Scanning Electronic Microscopy
Health Economy related to HRQL | At baseline, 9 weeks and at study completion 18 weeks (3 measurements)
  Questionnaire EQ-5D (scores transformed to Qaly) In- and out-patient costs for PICC/SVAP
Health Economy related to PICC and SVAP | Retrospective data assessment after study completion 18 weeks
  Device costs, maintenance costs (including complication cost), operation costs, staff costs retrieved from medical and economical records
Lived experience of complications | weekly, through study completion up to 18 weeks
  Structured diary filled by the participants regarding VAS, Visual Analog Scale
Lived experience of management of complications | weekly, through study completion up to 18 weeks
  Structured study specific diary filled by the participants regarding time management of device and complications.

CONTACTS AND LOCATIONS:
Overall Officials: Gunilla Björling, PhD, Study Chair — The Swedish Red Cross University College
Locations (1):
- Onkologiska kliniken, Karolinska University Hospital, Danderyd Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Data will be available 36 months after study completion.